CLINICAL TRIAL: NCT05480410
Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) on Pain and Quality of Life in Patients With Cancer Neuropathic Pain. Clinical Trial
Brief Title: Effectiveness of rTMS on Pain and Quality of Life in Patients With Cancer Neuropathic Pain. Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Universitaria Maria Cano (Other)
Responsible Party: Principal Investigator, Catalina Lopera Muñetón, Associate Professor, Fundacion Universitaria Maria Cano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 013008028-2021-311
Record Dates: First submitted 2022-06-10; First posted 2022-07-29 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain
Keywords: Transcranial Magnetic Stimulation, Repetitive; Neuropathic pain; Quality of life; Cancer
MeSH Terms: conditions — Neuralgia; Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A single group including patients with neuropathic oncological pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active intervention (Experimental): Patients will receive 20 sessions of transcranial magnetic stimulation applied with the MagVenture Mag Pro R20 equipment, these sessions will be held daily from Monday to Friday, lasting 20 minutes at an intensity of 81% with a motor threshold of 90 A/ns.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — rTMS is a minimal invasive technique which focus on the M1 cortex. It can stimulate the cortex by depolarizing superficial neurons. For this study we will use a MagVenture MagPro R20
  Other Names: rTMS

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Repetitive transcranial magnetic stimulation (rTMS) on pain and quality of life in patients with cancer neuropathic pain.

Although there are currently different therapeutic options for neuropathic pain, most are limited or restricted to pharmacotherapy. Transcranial magnetic stimulation (TMS) is a tool recently incorporated into neuroscience in the management of neuropathic cancer pain.

The study will include 10 patients with oncologic neuropathic pain who will receive 20 sessions of rTMS and the effect on pain and quality of life.

DETAILED DESCRIPTION:
Neuropathic pain is defined as pain caused by a primary lesion or transient dysfunction of the central or peripheral nervous system. In cancer, it is generated as a consequence of multiple factors such as: direct compression of nerve structures, post-surgical nerve injuries, and nerve injuries secondary to chemotherapy. At least 3.5 million people around the world suffer from this symptom associated with cancer; Of this population, 38% experience pain in all stages and 80% in advanced stages, negatively impacting quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuropathic pain of oncological origin
* Patients of legal age (18 years old)
* Patients using their cognitive faculties

Exclusion Criteria:

* Pregnancy
* History of negative reaction to TMS
* History of seizure, history of epilepsy stroke, brain surgery and cranial metal implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catalina Lopera, Msc, Principal Investigator — Fundacion Universitaria Maria Cano
Locations (1):
- CORTEX, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in oncological neuropathic pain. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will made accessible for up to 18 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact catalinaloperamuneton@fumc.edu.co

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Change of 20 rTMS Sessions on Pain
Description: Assessment of pain quantify by Visual analogue scale rated from 0-10, where 0 is the least pain and 10 the worst pain
Time Frame: Day 1 vs Day 20 vs 1st month follow up and vs 3rd month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention
Number analyzed (Participants) | 10
score on a scale
  Day 1 | 5.53 (1.27)
  Day 20 | 1.60 (1.47)
  1st month follow up | 1.97 (1.77)
  3rd month follow up | 3.48 (2.65)

2. Primary Outcome: Effect of Change of 20 rTMS Sessions on Pain and Functionality
Description: Assessment of pain severity and functionality quantify by brief pain inventory from 0-10, where 0 is the least pain and 10 the worst pain
Time Frame: Day 1 vs Day 20 vs 1st month follow up and vs 3th month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention
Number analyzed (Participants) | 10
score on a scale
  Day 1 Pain severity | 5.53 (1.27)
  Day 20 Pain severity | 1.60 (1.47)
  1st month follow up pain severity | 1.97 (1.77)
  3rd month follow up pain severity | 3.48 (2.65)
  Day 1 interference score | 5.75 (1.58)
  Day 20 interference score | 0.73 (1.03)
  1st month follow up interference score | 2.01 (1.59)
  3rd month follow up interference score | 3.30 (2.27)

3. Secondary Outcome: Effect of Change of 20 rTMS Sessions on Quality of Life
Description: Assessment of Quality of life, measured by Functional Assessment of cancer Therapy (FACT-GOG- NTX 13) (0-100) higher number means a better quality of life
Time Frame: Day 1 vs Day 20 vs 1st month follow up and vs 3rd month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention
Number analyzed (Participants) | 10
score on a scale
  Day 1 FACT Total score | 68.90 (7.62)
  Day 20 FACT total score | 91.00 (9.23)
  1st month follow up FACT total score | 85.10 (15.08)
  3rd month follow up FACT total score | 79.50 (16.90)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Active Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Intervention (N=10)
drowsiness (Nervous system disorders) | 1 (1)
Mild headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations in the interpretation of our results include the small sample size of this pilot study, the lack of a sham stimulation group. Future research with longer follow up could support the inclusion of rTMS as a therapeutic option for comprehensive oncology rehabilitation programs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05480410/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT05480410/SAP_001.pdf